CLINICAL TRIAL: NCT03669328
Title: Evaluation of Pain and Postoperative Nausea Vomiting Incidence in Outpatient Surgery at IUCT-Oncopole Hospital
Status: Completed | Type: Observational
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Other Study IDs: 16HLGENF01
Record Dates: First submitted 2018-08-30; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Anesthesia; Cancer; Surgery
Keywords: Surgery; cancer; anesthesia; pain; outcome patient; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Neoplasms; Pain; Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: patients of 2016, June with locoregional anesthesia
  Interventions: Procedure: locoregional anesthesia
- Group 2: patients of 2018, June with locoregional anesthesia
  Interventions: Procedure: locoregional anesthesia

INTERVENTIONS:
Procedure: locoregional anesthesia — Both groups received locoregional anesthesias

SUMMARY:
The effectiveness of the analgesic and anti-nausea prevention techniques of the investigators justifies being evaluated regularly in order to adapt the management strategy to the specificities of each surgical act.

A first evaluation took place in June 2016 and allowed to identify a category of patients (partial breast surgery with or without axillary gesture) not benefiting from an ideal algological management because justifying in 30% of the cases of a level 3 analgesic remedy in the postoperative recovery room. This use of morphine results in a significant incidence of postoperative nausea and prolonged recovery time before return home harmful to the patient.

With their experience in locoregional anesthesia technique in complete breast surgery (total mastectomy) and aware of the effectiveness of this type of anesthesia on the management of immediate and chronic pain, the investigators have extended their indications of ALR to partial breast surgery in ambulatory.

DETAILED DESCRIPTION:
During the anesthesia consultation, the risk of postoperative nausea and vomiting (PONV) is evaluated by the Apfel score (Apfel CC, Anesthesiology 1999) and a preventive strategy correlated to this score is then determined. An order including anti-emetics and analgesics is given to the patient for the return home after the outpatient surgery.

On the day of the outpatient surgery, patients receive in the operating room the prevention of PONV according to their level of risk (according to the recommendations of the Société Française d'Anesthésie et de Réanimation - SFAR 2008 and Guidelines 2014) and analgesics including a level II and NSAIDs (in the absence of contraindication).

All patients underwent general anaesthesia with sufentanil and propofol. Mechanical ventilation was performed with laryngeal mask. A echoguided regional anesthesia was performed by injection of 20 ml of ropivacaine 3.75 mg/ml above and under the serratus muscle as described by Blanco and al (ref 3)" In the postoperative recovery room, PONV is treated if necessary by an anti-emetic class different from those used in the block. In postoperative pain with EVA> 3, morphine titration is performed as recommended.

Patients are then monitored in an outpatient surgery unit until they have a home-based return capability assessed by the CHUNG score, including the level of pain (moderate and well relieved), the absence of persistent nausea, and the ability to ambulation.

All outpatient surgery patients are called the day after their return home to ensure the absence of complications according to the regulatory procedure related to outpatient anesthesia.

As part of this evaluation, information on the level of pain at rest and mobility, as well as the frequency of PONV are also recorded and this follow-up is repeated in D2 and D3 after the intervention.

This information is then correlated with the type of anesthesia performed, the surgical procedure as well as the analgesic strategy (ALR) and the antinausea strategy performed.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted for ambulatory surgery under general anesthesia
* patients admitted during the period from 01 to 30 June 2016 or during the period from 18 to 5 July 2018

Exclusion Criteria:

* Patient neither French nor English,
* Patient refusing to participate in this study
* Minor patients were excluded to ensure the homogeneity of the surveyed population (satisfaction of minors not meeting the same characteristics as that of adults)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During the period from 01 to 30 June 2016, all patients admitted for ambulatory surgery under general anesthesia were included in this prospective "before-after" study.
  To have two perfectly comparable populations, we chose to reassess all patients in outpatient surgery combined, on the second period (18 to 5 July 2018), even if our changes of care only concerns breast.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain after surgery by Simple Verbal Evaluation | 1 day (the day of the surgery)
  Pain level in post-operative room measured by Simple Verbal Evaluation. The simple verbal scale or Keele scale has 5 qualifiers to describe the intensity of the pain, each descriptor is associated with a numerical value. 0 = no pain, 1 = poor, 2 = moderate, 3 = intense, 4 = atrocious.
  The goal of management is to achieve pain values below 3 (low to moderate).

SECONDARY OUTCOMES:
Incidence of postopérative nausea and vomiting after prevention strategy guided by Apfel score risk | 1 day before surgery
  The risk of postoperative nausea and vomiting (PONV) is evaluated by the Apfel score and a preventive strategy correlated to this score is then determined. An order including anti-emetics and analgesics is given to the patient for the return home after the outpatient surgery. The Apfel score includes four variables (Female sex, History of motion sickness or postoperative nausea and vomiting, Nonsmoker, Postoperative opioid treatment is planned) and assigns one point for each.
Medical procedure characteristics | 1 day (the day of the surgery)
  The type of anesthesia performed, the surgical procedure as well as the analgesic strategy (ALR) and the antinausea strategy performed.
Evaluation of pain after surgery by Opioid requirements | 3 days (from surgery to 3 days after)
  Pain level in post-operative room measured and opioid requirement if important pain persists. The scale used is the "visual analogue scale ". If EVA> 3 titration with morphine 1 mg per 1 mg is performed in the recovery room until an EVA <3 is obtained. The dose of morphine in mg necessary to achieve this objective is collected.
Evaluation of home-based return capability by CHUNG score | 1 day (just after the surgery)
  Patients are then monitored in an outpatient surgery unit until they have a home-based return capability assessed by the CHUNG score, including the level of pain (moderate and well relieved), the absence of persistent nausea, and the ability to ambulation.Points are assigned to six variables : level of consciousness, physical activity, hemodynamic stability, oxygen saturation, pain, emetic symptoms. A score of 9 or 10 is needed to allow the patient to leave the hospital.
Evaluation of pain at home after surgery at mobility by EVA during the first 3 days | 3 days (from surgery to 3 days after)
  Pain level (Analogic Visual Evaluation EVA) on the first 3 days after surgery at mobility. The EVA is a numeric scale of pain. The patient must estimate his pain level from 0 (no pain) to 10 (the most unsustainable pain ever experienced). The question asked by phone is "between 0 no pain and 10 excruciating pain, where would you place your pain on this scale?" This scale is validated by the entire scientific community as the most sensitive and above all the most reproducible and can be obtained by phone.
  an acceptable pain is <3 therefore mild to moderate.
Evaluation of pain at home after surgery at rest by EVA during the first 3 days | 3 days (from surgery to 3 days after)
  Pain level (Analogic Visual Evaluation EVA) on the first 3 days after surgery, at rest. The EVA is a numeric scale of pain. The patient must estimate his pain level from 0 (no pain) to 10 (the most unsustainable pain ever experienced). The question asked by phone is "between 0 no pain and 10 excruciating pain, where would you place your pain on this scale?" This scale is validated by the entire scientific community as the most sensitive and above all the most reproducible and can be obtained by phone.
  an acceptable pain is <3 therefore mild to moderate.
Evaluation of sleep quality | 3 days (from surgery to 3 days after)
  Sleep quality (wake up by pain or not during the night) during the 3 days after surgery. Patient is asked to answer yes or not to the question : Have you been awakened by pain during the night" during first 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Amel Daboussi, PhD, Principal Investigator — Institut Claudius Regaud
Locations (1):
- Institut Claudius Regaud, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Result] Fuzier R, Puel F, Izard P, Sommet A, Pierre S. Prospective cohort study assessing chronic pain in patients following minor surgery for breast cancer. J Anesth. 2017 Apr;31(2):246-254. doi: 10.1007/s00540-016-2288-9. Epub 2016 Nov 24. PMID 27885426
- [Result] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Result] Bouhassira D, Attal N, Alchaar H, Boureau F, Brochet B, Bruxelle J, Cunin G, Fermanian J, Ginies P, Grun-Overdyking A, Jafari-Schluep H, Lanteri-Minet M, Laurent B, Mick G, Serrie A, Valade D, Vicaut E. Comparison of pain syndromes associated with nervous or somatic lesions and development of a new neuropathic pain diagnostic questionnaire (DN4). Pain. 2005 Mar;114(1-2):29-36. doi: 10.1016/j.pain.2004.12.010. Epub 2005 Jan 26. PMID 15733628
- [Result] Kumar SP. Utilization of brief pain inventory as an assessment tool for pain in patients with cancer: a focused review. Indian J Palliat Care. 2011 May;17(2):108-15. doi: 10.4103/0973-1075.84531. PMID 21976850